CLINICAL TRIAL: NCT01639833
Title: A Premarket, Prospective, Randomized, Single-Blind Study to Compare the Veriset™ Hemostatic Patch to TachoSil® as an Adjunct to Hemostasis in Subjects Undergoing Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: COVEUCV0140
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Surgical Procedures; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Veriset Hemostatic Patch (Experimental): Topical Hemostat
  Interventions: Device: Veriset Hemostatic Patch
- TachoSil® (Active Comparator): Topical Hemostat
  Interventions: Device: TachoSil®

INTERVENTIONS:
Device: Veriset Hemostatic Patch — Topical hemostat
  Arms: Veriset Hemostatic Patch
Device: TachoSil® — Topical Hemostat
  Arms: TachoSil®

SUMMARY:
The objective of this study is to assess the safety and effectiveness of Veriset™ Hemostatic Patch in cardiovascular procedures by comparing Veriset™ Hemostatic Patch to TachoSil® in subjects undergoing open cardiovascular surgery involving the aorta (e.g., aortic valve replacement (AVR), David procedure, Bentall procedure, abdominal aortic aneurysm repair, etc.), or CABG.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Subject is ≥18 years of age.
* Subject is scheduled for surgery involving the aorta (e.g., aortic valve replacement (AVR), David procedure, Bentall procedure, abdominal aortic aneurysm repair, etc.), or coronary artery bypass graft (CABG) where a topical hemostatic agent would be used to control bleeding via an open approach.
* Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.
* Subject is undergoing emergency surgery, i.e. lifesaving procedures performed where patient is in imminent danger of death.
* Subject has a history of allergic reactions after application of human fibrinogen, human thrombin and/or collagen of any origin.
* Subject is pregnant (documented by a positive pregnancy test) or is actively breast-feeding.
* Subject has an estimated life expectancy of less than 6 months.
* Subject is unwilling to receive blood products.
* Subject is scheduled for another planned cardiovascular surgery, and subsequent surgery would jeopardize previous application of study treatment.
* The subject has participated in another investigational drug or device research study within 30 days of enrollment.

Exclusion Criteria:

* Subject has an appropriate Target Bleeding Site (TBS) defined as an area of bleeding on the aorta or coronary vessels where hemostasis by conventional methods is ineffective or impractical, and thus necessitates the use of a topical hemostatic agent.
* TBS Bleeding is Type 2 (Oozing/Mild) or 3 (Moderate).
* It is possible to hold pressure on Veriset™ Hemostatic Patch or TachoSil® for at least 3 minutes.
* Incidental finding of any other pre-operative exclusion criteria
* Subject does not have an appropriate TBS.
* TBS Bleeding Assessment is Type 1 (No bleeding) or 4 (Severe/Surgical/Life Threatening).
* Subject has an active local infection at the surgical site.
* Investigator determines that participation in the study may jeopardize the safety or welfare of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Glineur, MD, Principal Investigator — Clinique St-Luc Bouge, Namur, Belgium
Locations (12):
- Belgium (6):
  - Bonheiden
  - St Luc Hospital, Brussels
  - UZ Brussels, Brussels
  - Genk
  - Hassalt
  - Leuven
- Germany (5):
  - Dresden
  - Freiburg im Breisgau
  - Hamburg
  - Leipzig
  - Munich
- Riga, Latvia

RESULTS

PARTICIPANT FLOW:
Groups:
- Veriset™ Hemostatic Patch: Topical Hemostat
  Veriset™ Hemostatic Patch: Topical hemostat
Period: Overall Study
Arm/Group | Veriset™ Hemostatic Patch | TachoSil®
Started | 45 | 45
Completed | 39 | 41
Not Completed | 6 | 4
Not completed — Death | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veriset™ Hemostatic Patch | TachoSil® | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (12.2) | 66.7 (13.4) | 67.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 29 | 32 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 44 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 171.3 (9.1) | 170.8 (10.4) | 171.1 (9.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 81.67 (14.27) | 81.96 (17.27) | 81.82 (15.75)

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis (TTH)
Description: Time to Hemostasis (TTH) at the target bleeding site (TBS) following treatment (Veriset™ Hemostatic Patch or Control).
Time Frame: Day 0
Population: The Per Protocol (PP) population was used for the primary analysis of the primary effectiveness endpoint for the non-inferiority test.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Veriset™ Hemostatic Patch | TachoSil®
Number analyzed (Participants) | 41 | 45
minutes | 1.50 [1.50 to 2.00] | 3.00 [NA to NA] — Confidence interval was calculated using the Brookmeyer and Crowley method. 91% of TachoSil® patients achieved hemostasis at 3 minutes and no patient had hemostasis before 3 minutes. The confidence interval of the median time cannot be estimated.

2. Secondary Outcome: Hemostasis at All Treated Bleeding Sites Within 3 Minutes
Description: The proportion of subjects achieving hemostasis at all treated bleeding sites within 3 minutes of device application.
Time Frame: Day 0
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Veriset™ Hemostatic Patch | TachoSil®
Number analyzed (Participants) | 41 | 45
percentage of participants | 87.8 [77.8 to 97.8] | 91.1 [82.8 to 99.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 90 day follow-up visit.
Description: All adverse events were reported, regardless of relationship to study device.
Arm/Group | Veriset™ Hemostatic Patch | TachoSil®
Serious Adverse Events (participants affected / at risk) | 13/44 | 11/45
Other Adverse Events (participants affected / at risk) | 23/44 | 21/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Veriset™ Hemostatic Patch (N=44) | TachoSil® (N=45)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular failure (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Cardiac output decreased (Investigations) | 1 | 0
Hemianopia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Veriset™ Hemostatic Patch (N=44) | TachoSil® (N=45)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Atrial Fibrillation (Cardiac disorders) | 13 | 10
Urinary tract infection (Infections and infestations) | 3 | 0
Delirium (Psychiatric disorders) | 3 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Pericardial effusion (Cardiac disorders) | 0 | 4
Renal failure (Renal and urinary disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No